CLINICAL TRIAL: NCT07173972
Title: PROSARC-2. Dose-escalated, Hypofractionated, Definitive Proton Radiotherapy for Patients With Inoperable Soft Tissue Sarcoma. A Single-arm, Multicenter, Phase II Clinical Trial.
Brief Title: Dose-escalated, Hypofractionated, Definitive Proton Radiotherapy for Patients With Inoperable Soft Tissue Sarcoma.
Acronym: PROSARC-2
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: Haukeland University Hospital (Other); St. Olavs Hospital (Other); University Hospital of North Norway (Other)
Responsible Party: Principal Investigator, Ivar Hompland, Senior Consultant, MD, PhD, Oslo University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 916024
Record Dates: First submitted 2025-09-08; First posted 2025-09-15 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Soft Tissue Sarcoma (STS); Soft Tissue Sarcoma Adult; Soft Tissue Sarcoma of the Trunk and Extremities; Synovial Sarcomas; Undifferentiated Pleomorphic Sarcoma (UPS); Myxofibrosarcoma; Leiomyosarcoma (LMS); Pleomorphic Liposarcoma; Pleomorphic Rhabdomyosarcoma; Liposarcoma
Keywords: soft tissue sarcoma; proton radiotherapy; inoperable soft tissue sarcoma
MeSH Terms: conditions — Sarcoma; Sarcoma, Synovial; Histiocytoma, Malignant Fibrous; Dermatofibrosarcoma; Leiomyosarcoma; Liposarcoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Inoperable soft tissue sarcoma (Experimental)
  Interventions: Radiation: Definitive radiotherapy

INTERVENTIONS:
Radiation: Definitive radiotherapy — The prescribed dose is 56 Gray (Gy) in 16 fractions over 4 weeks (14 Gy per week) with a maximum dose-escalation to the tumor core of 80 Gy (5 Gy per fraction).

SUMMARY:
The purpose of the study is to study if dose escalated proton radiotherapy can improve local controll for patients with inoperable soft tissue sarcomas. The standard treatment is photon-based radiation. By using proton radiotherapy instead, the hypothesis is that the dose can be increased to enhance treatment effectiveness without increasing side effects.

The planned radiation dose is 56 Gy in 16 fractions (treatments) over 4 weeks (4 fractions per week), with a maximum dose escalation centrally in the tumor up to 80 Gy (5 Gy per fraction).

At the same time, the study will investigate biomarkers that can predict treatment response, including changes in the tumor's genetic material (DNA), measurements of various molecules in the bloodstream, and the tumor's appearance on MRI scans.

The primary endpoint is local control after 2 years, meaning that the treated tumor has not grown during this period. Secondary endpoints include overall survival, progression-free survival, radiological response rates, side effects, and quality of life.

The study will be conducted in Norway, with a planned inclusion of 40 patients.

DETAILED DESCRIPTION:
The objective of the PROSARC-2 trial is to investigate whether dose-escalated hypofractionated, definitive, proton beam therapy (PBT) can result in better local control in soft tissue sarcoma (STS). PROSARC-2 is a single arm, open-label, multicenter phase II clinical trial initiated at the Department of Oncology, Oslo University Hospital (OUS). The main inclusion criterion is patients with inoperable soft tissue sarcoma. The primary endpoint is 2-year local progression-free survival (LPFS). We expect to include 40 patients over three years and all patients will be followed for up to five years. All the sarcoma centers in Norway participate in the study: OUS; Haukeland University Hospital (HUH); St Olavs Hospital (SOH) and University Hospital of North-Norway (UNN). The indication for definitive radiotherapy (RT) will be decided in the sarcoma multidisciplinary (MDT) meeting at each center. A weekly/biweekly national sarcoma RT meeting will make the decision whether hypofractionated, dose-escalated PBT will be feasible after a careful clinical evaluation. For included patients PBT will be given at OUS and HUH. The prescribed dose is 56 Gray (Gy) in 16 fractions over 4 weeks (14 Gy per week) with a maximum dose-escalation to the tumor core of 80 Gy (5 Gy per fraction).

The PROSARC-2 trial includes translational radiomic research, where we aim to elucidate underlying mechanisms related to RT effect. To facilitate future biomarker studies for personalized therapy we will collect excess tumor tissue, whole blood, plasma and serum.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18 years of age at the time of informed consent.
2. Histological diagnosis of soft tissue sarcoma including gastrointestinal stromal tumor (GIST).
3. Measurable disease according to RECIST v1.1.
4. Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1 or 2
5. For patients with metastatic disease a life-expectancy greater than 2 years should be expected.
6. Before patient registration, written informed consent must be given according to national and local regulations.
7. Ability to fill in patient questionnaires and comply with study procedures, including travelling to Bergen or Oslo for Proton Beam radiotherapy.

Exclusion Criteria:

1. Patients with a prior or concurrent malignant disease whose natural history or treatment have the potential to interfere with the safety or efficacy assessment of this clinical trial are not eligible. Patients with a history of breast cancer, requiring continued hormonal treatment (e.g. anti-estrogen or an aromatase inhibitor) may be included. Patients with a history of prostate cancer, requiring continued support with luteinizing hormone releasing hormone (LHRH) agonists, with or without androgens, may be included.
2. Previous radiotherapy to the tumor site.
3. Patients with pacemakers and/or implanted defibrillators.
4. Patients not able to give an informed consent or comply with study regulations as deemed by study investigator.
5. Administration of systemic cancer therapy (i.e. chemotherapy, targeted therapy or immune therapy) within 14 days prior to the first fraction of radiotherapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-01-26 (Actual); Primary Completion 2029-01-26 (Estimated); Study Completion 2035-11-01 (Estimated)

PRIMARY OUTCOMES:
Local progression-free survival | 2 Year
  Local progression-free survival is measured from the date of start of study treatment until date of local progression of the tumor that has undergone proton beam radiotherapy evaluated using RECIST v1.1 or date of death of any cause, whichever occurs first.

SECONDARY OUTCOMES:
Progression-free survival | Up to five years after radiation therapy
  Progression-free survival is measured from the date of start of study treatment until date of progressive disease (local and/or distant) as evaluated using RECIST v1.1 or date of death of any cause, whichever occurs first.
Overall survival | Up to five years after radiation therapy.
  Overall survival is measured from the date of start of study treatment until date of death of any cause.
Overall response rate, defined as partial or complete response using RECIST v1.1 | Up to five years after radiation therapy.
  Radiological response will be assessed using MRI and/or CT of the primary tumor.
Health-related quality of life | Up to five years after radiation therapy.
  Change from baseline in EORTC QLQ-C30 scores.
To assess acute and late toxicity | Up to five years after radiation therapy.
  Treatment-related toxicity during treatment and follow-up using CTCAE v5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Ivar Hompland, MD, PhD, Principal Investigator — Oslo University Hospital; Kjetil Boye, MD, PhD, Study Director — Oslo University Hospital
Locations (2):
- Norway (2):
  - Haukeland University Hospital, Bergen
  - Oslo University Hospital, Oslo

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR